CLINICAL TRIAL: NCT04774848
Title: High Frequency Oscillatory Ventilation Versus High Frequency Jet Ventilation as Initial Mode of Ventilation for Congenital Diaphragmatic Hernia
Brief Title: High Frequency Oscillatory Ventilation Versus High Frequency Jet Ventilation for Congenital Diaphragmatic Hernia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Michelle Yang, Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 133683
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-01

CONDITIONS: Congenital Diaphragmatic Hernia
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Intervention Model Description: Infants stratified by presence of intrathoracic liver (yes/no) and are randomized to either high frequency jet ventilator or high frequency oscillating ventilator in a sequential 1:1 manner
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- High Frequency Jet Ventilation (HFJV) with intrathoracic liver (Active Comparator): Babies known to have the presence of the liver in the intrathoracic space will be placed on the HFJV at delivery or as soon as possible after consent. During analysis, these babies will be compared to babies with intrathoracic liver and randomized to high frequency oscillating ventilator.
  Interventions: Device: High Frequency Jet Ventilator
- High Frequency Jet Ventilation (HFJV) without intrathoracic liver (Active Comparator): Babies who do not have any liver in the intrathoracic space will be placed on the HFJV at delivery or as soon as possible after consent. During analysis, these babies will be compared to babies without intrathoracic liver and randomized to high frequency oscillating ventilator.
  Interventions: Device: High Frequency Jet Ventilator
- High Frequency Oscillatory Ventilation (HFOV) with intrathoracic liver (Active Comparator): Babies known to have the presence of the liver in the intrathoracic space will be placed on the HFOV at delivery or as soon as possible after consent. During analysis, these babies will be compared to babies with intrathoracic liver and randomized to HFJV.
  Interventions: Device: High Frequency Oscillatory Ventilator
- High Frequency Oscillatory Ventilation (HFOV) without intrathoracic liver (Active Comparator): Babies who do not have any liver in the intrathoracic space will be placed on the HFOV at delivery or as soon as possible after consent. During analysis, these babies will be compared to babies without intrathoracic liver and randomized to HFJV.
  Interventions: Device: High Frequency Oscillatory Ventilator

INTERVENTIONS:
Device: High Frequency Jet Ventilator — HFJV provides short bursts of gas into the respiratory circuit at a rate of 240 to 600/min (4 to 11 Hz) and expiration is passive. It is used in conjunction with a conventional ventilator which provides positive end expiratory pressure (PEEP) and can also provide occasional sigh breaths.
  Arms: High Frequency Jet Ventilation (HFJV) with intrathoracic liver; High Frequency Jet Ventilation (HFJV) without intrathoracic liver
Device: High Frequency Oscillatory Ventilator — HFOV uses a piston diaphragm to generate alternating positive and negative pressure changes to give breaths of 300 to 900/min (5-15 Hz) given over a set mean airway pressure. Both inhalation and exhalation are active.
  Arms: High Frequency Oscillatory Ventilation (HFOV) with intrathoracic liver; High Frequency Oscillatory Ventilation (HFOV) without intrathoracic liver

SUMMARY:
The purpose of this study is to conduct a prospective study of all congenital diaphragmatic hernia (CDH) neonates managed at the University of Utah newborn intensive care unit (NICU) and Primary Children's Hospital NICU that required mechanical ventilation at birth. As both high frequency jet ventilation (HFJV) and high frequency oscillatory ventilation (HFOV) are standard approaches to ventilatory support of all neonates including CDH, CDH infants will be randomized at the time of birth or admission to either HFJV or HFOV as initial ventilator mode, stratified by position of the liver in the abdomen or thorax (if known) by 24 hours of age. Measures of oxygenation, ventilation and hemodynamics of the CDH cohort managed on HFOV compared to those on HFJV.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to either the University of Utah and/or Primary Children's Hospital NICU within 24 hours of birth
2. Requiring mechanical ventilation
3. Umbilical arterial line or peripheral arterial line in place
4. Obtained signed consent
5. Infant is ≤ 24 hours of age

Exclusion Criteria:

1. Severe anomaly

   1. Chromosomal abnormalities
   2. Major congenital anomalies, including cardiac, central nervous system and syndromes
2. Post-natal diagnosis > 24 hours of life
3. Unable to obtain consent for participation
4. Unable to randomize within 24 hours of life

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2020-12-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-28 (Estimated)

PRIMARY OUTCOMES:
Oxygenation Index (OI) at 24 hours of age | 24 hours of age
  The OI will be measured at 24 hours of age using a standard of care arterial blood gas and oxygen settings. These measurements will then be compared between the stratified groups

SECONDARY OUTCOMES:
PF ratio (PaO2/FiO2) measurements | up to one week
  These measurements will be determined at multiple time points for the first week of life. These measurements will be compared between groups.
PF-PCO2 (PaO2/FiO2-PaCO2) measurements | up to one week
  These measurements will be determined at multiple time points for the first week of life. These measurements will be compared between groups.
PaCO2 measurements | up to one week
  These measurements will be determined at multiple time points for the first week of life. These measurements will be compared between groups.
Number of babies who received inhaled nitric oxide (iNO) | up to one week
  the number of babies who received treatment of iNO will be compared amongst the different groups

OTHER OUTCOMES:
Number of babies who survive to discharge | up to one year
  the number of babies who survive and are discharged will be compared amongst the groups
Number of babies who required extracorporeal membrane oxygenation (ECMO) | up to one year
  the number of babies who required ECMO will be compared amongst the groups
Number of days on mechanical ventilation | up to one year
  the number of days each baby required intubation and mechanical ventilation by any type will be compared amongst the groups

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Yang, MD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Primary Children's Hospital, Salt Lake City, Utah
  - University Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No